CLINICAL TRIAL: NCT05911321
Title: Study of Isatuximab Plus Pomalidomide and Dexamethasone in Highly Toxicity-vulnerable Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Isa-Pom-Dex in Elderly/Frail Subjects With RRMM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2119
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma; Relapse; Refractory; Aging; Co-morbidity
Keywords: Pomalidomide; Isatuximab; Dexamethasone; low dose
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — isatuximab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Subjects with relapsed or refractory multiple myeloma receiving the study treatment.
  Interventions: Drug: Isatuximab; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — Pharmaceutical form: Solution for infusion. Route of administration: Intravenous 10 mg/kg will be administered intravenously once weekly during cycle 1 and every other week during each subsequent cycle.
Drug: Pomalidomide — Pharmaceutical form: Pill for oral use. Route of administration: 3 mg Pomalidomide 3 mg pill will be taken by mouth once daily on days 1-21 of each 28-day cycle.
Drug: Dexamethasone — Pharmaceutical form: Tablet for oral use Route of administration: Pill for oral use. Dexamethasone 20 mg tablet will be taken by mouth once per week.

SUMMARY:
This research study aims to evaluate the safety and effectiveness of the combination of isatuximab, pomalidomide, and dexamethasone (Isa-Pd) for the treatment of relapsed or refractory multiple myeloma (RRMM), which refers to multiple myeloma that has returned or has not responded to prior treatment. The study will specifically investigate the impact of administering lower-than-standard doses of pomalidomide and dexamethasone. Using lower doses of pomalidomide and dexamethasone in this setting has not been approved by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
This study aims to address the challenges faced in selecting appropriate therapy for elderly or highly toxicity-vulnerable patients who are poor candidates for standard (full-dose) chemotherapy regimens. Traditional clinical trials often exclude these patients, limiting the generalizability of available data. This single-arm multicenter phase II study will enroll 49 older and/or toxicity-vulnerable patients with RRMM. The study will evaluate the safety and effectiveness of isatuximab when used in combination with pomalidomide and dexamethasone at lower than standard doses. The primary objective is to estimate the overall response rate (ORR), while secondary objectives include the estimation of additional measures of response, as well as measures of toxicity and tolerability. All participants in the trial will also be evaluated by Cancer and Aging Research Group Geriatric Assessments (CARG-GA) and patient- reported outcome (PRO) measures of quality of life (QOL). Biomarkers of aging and frailty will also be studied.

Duration of therapy:

The duration of study participation will depend on the response to the treatment. In the absence of treatment delays due to adverse events, treatment with Isa-Pd will generally continue until disease progression, unacceptable side effects, other illness or condition that prevents further study treatment, or a subject's decision to withdraw from the study. On average, subjects will most likely be treated for approximately 10 months on this study.

Duration of Follow-Up:

All participants, including those withdrawn for adverse events (AEs) will be followed after removal from study treatment until death or full subject withdrawal from the study for other reasons. Participants removed from the study treatment for unacceptable AEs will be followed for resolution or stabilization of the AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained to participate in the study and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information (PHI). Consent must be obtained before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. Age ≥ 18 years at the time of consent.
3. Documented symptomatic multiple myeloma that has previously responded to therapy (partial response or better) and is relapsed or relapsed and refractory to the last line of therapy.
4. Patients must also be refractory to at least one prior line of therapy that includes an IMiD and/or a PI, and should have received at least 2 cycles of that regimen to be evaluable for refractoriness .
5. If previously treated with an anti-CD38 containing regimen, the subject must have achieved at least a PR to that line of therapy and must not have received an anti- CD38 mAb for at least 6 months prior to enrollment.
6. Willing and able to adhere to the study visit schedule and other protocol requirements based on the judgement of the investigator.
7. Predicted high risk for severe toxicity from intensive regimens for RRMM, such as standard (full-dose) DPD, DVD, KPD, KRD, Ixa-PD, or Elo-PD as each regimen was published (such regimens often use, for example, twice-weekly bortezomib at 1.3 mg/m2, lenalidomide at 25 mg, or pomalidomide 4 mg). High-risk is defined as one of the following:

A. Score ≥ 2 (indicating "frail") on the International Myeloma Working Group instrument (IMWG; Palumbo et al. [Blood 2015]) B.KPS ≤ 70

C. Not meeting criteria A or B above but felt by treating clinician to not be a candidate for a standard full-dose regimen on account of one of the following:

i) History of clinically significant non-hematologic grade ≥3 (NCI CTCAE, version 5.0) toxicity attributed to prior anticancer therapy ii) History of requiring dose-reduction of at least two separate anticancer drugs during prior therapy for multiple myeloma.

Exclusion Criteria:

All subjects meeting any of the listed exclusion criteria at baseline with be excluded from study participation.

1. Anti-myeloma treatment within 2 weeks of cycle 1 day 1
2. Prior treatment with pomalidomide
3. Any monoclonal antibody therapy within the previous 30-days
4. Anti-CD38 monoclonal antibody therapy within the previous 6 months
5. Autologous stem cell transplantation within 12 weeks of day 1 of cycle 1
6. Subjects felt to not be candidates by treating physician for any systemic therapy due to excessive comorbidities, frailty, impaired performance status, or other severe limitations. Such limitations can be conceptualized generally as making subjects exceedingly high risk for any systemic treatment. These limitations often stem from medical comorbidities unrelated to MM and they are hence unlikely to improve with MM therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2028-03-26 (Estimated)

PRIMARY OUTCOMES:
Overall response Rate (ORR) | Up to 12 weeks
  ORR is defined as a partial response or better (≥PR) to study therapy at any time, based on International Myeloma Working Group (IMWG) criteria.
  Complete response (CR): Negative immunofixation of serum and urine, disappearance of soft tissue plasmacytomas, and <5% plasma cells in bone marrow (BM). Stringent complete response(sCR): CR plus normal free light chains (FLC) ratio and absence of clonal plasma cells in BM biopsy. Very good partial response (VGPR):-Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M component plus urine M component <100/24h. Partial response (PR) ≥50% reduction of serum M-protein & reduction in 24-hour (24h) urinary M-protein by ≥90% or to <200 mg/24h and if present at baseline, a ≥ 50% reduction in the size soft tissue plasmacytomas.

SECONDARY OUTCOMES:
Treatment related adverse events rate | Up to 12 weeks
  All treatment-related adverse events as defined by changes from baseline utilizing National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0.
  NCI-CTCAE is a descriptive terminology utilized for AE reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Treatment failure-free survival (TFFS) | Up to 3 years
  TFFS is defined as the time start from the first day of study therapy until discontinuation for any reason, including disease progression, toxicity, or death.
  Progressive disease: Serum M-protein: absolute increase must be ≥ 0.5 g/dL, ≥ 1 g/dL if the lowest M component was ≥ 5 g/dL; absolute Urine M-protein increase≥ 200 mg/24 h). In patients without measurable serum and urine M-protein levels, the difference between involved and uninvolved FLC levels must be > 10 mg/dL; without measurable involved FLC levels, bone marrow plasma cell percentage irrespective of baseline status Appearance of a new lesion(s), ≥ 50% increase from nadir > 1 lesion, or ≥ 50% increase in the longest diameter of a previous lesion >1 cm in short axis;≥ 50% increase e in circulating plasma cells (minimum of 200 cells per μL) if this is the only measure of disease.
Maximum depth of response | Up to 12 weeks
  Maximum depth of response includes the summation of minimal response (MR), partial response (PR), very good partial response (VGPR), complete response (CR), and stringent complete response (sCR) based on IMWG criteria. Minimal response(MR): ≥ 25% but ≤ 49% reduction of serum M-protein and reduction in 24-h urine M-protein by 50-89%, if present at baseline, a ≥ 50% reduction in the size of soft tissue plasmacytomas is also required. PR, VGPR, CR, and sCR were defined above.
Clinical benefit rate (CBR) | Up to 12 weeks
  CBR is defined as a partial response or better (≥PR) + minimal response (MR) rate based on International Myeloma Working Group (IMWG) criteria.
Bone marrow minimal residual disease (MRD) negativity | Up to 12 weeks
  Bone marrow minimal residual disease (MRD) negativity will be defined as the ratio of subjects who achieved MRD to all subjects. MRD negativity will be assessed by next-generation sequencing with a minimum sensitivity of 1x10-5.
Time to first response | Up to 12 weeks
  Time to first response is defined as the time from the first study treatment to the achievement of PR or better as defined by IMWG criteria.
Time to best response | Up to 12 weeks
  Time to best response is defined as the time from the first study treatment to the achievement of best response (PR, VGPR, CR, or sCR) based on IMWG criteria.
Duration of response | Up to 3 years
  Duration of response is defined as the time from the achievement of PR or better until progressive disease (PD) based on IMWG criteria. Subjects will be censored if they die of anything other than myeloma.
Progression-free survival (PFS) | Up to 3 years
  PFS is defined as the time from the first study treatment until confirmed PD based on IMWG criteria or death from any cause, whichever comes first.
Median time to next treatment (TTNT) | Up to 3 years
  Median time to next treatment (TTNT) is defined as the time from the start of the study treatment to the next type of Multiple Myeloma treatment or death from any cause, whichever occurs first.
Overall survival | Up to 3 years
  Overall survival is defined as the time from the first study treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Eben I Lichtman, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials